CLINICAL TRIAL: NCT04531566
Title: Preterm Functional Early Enteral Development (FEED) Trial on Respiratory Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Ashley N Morin, Fellow, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-20-0741
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Premature Birth
Keywords: Prematurity; Oral Skills; Nasal CPAP oral feeds; HFNC oral feeds
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Feed Intervention Group (Experimental)
  Interventions: Dietary Supplement: Oral Feed
- Usual care (Active Comparator)
  Interventions: Dietary Supplement: Usual care

INTERVENTIONS:
Dietary Supplement: Oral Feed — Infant will be seen by occupational therapist (OT) twice a week and assessed for oral cues. If infant shows oral cues then the occupational therapist will proceed with feeding strategies. Oral feeding strategies include pacifier dips, open nipple trials with syringe controlled bolus size (1-4mls) and po trials up to 10mls.
  Arms: Oral Feed Intervention Group
Dietary Supplement: Usual care — Infants will not start oral feeds until on HFNC 2 Litres or less. Oral feeds will be started on the discretion of the physician.
  Arms: Usual care

SUMMARY:
The purpose of this study is to demonstrate that allowing infants that require high flow nasal cannula (HFNC)/Continuous positive airway pressure (CPAP) to orally feed if demonstrating oral cues will achieve full oral feeds faster.

ELIGIBILITY:
Inclusion Criteria:

* infants that require greater than 2 litres per minute (LPM) high flow nasal canula or CPAP with a max setting of 6cm H20 FiO2 30% or less for at least 72 hours or more
* Tolerating enteral feeds of 120 ml/kg/day

Exclusion Criteria:

* Major congenital anomalies (pulmonary malformations, airway malformations, craniofacial defects, major congenital heart disease, combined pulmonary intestinal malformations)
* Metabolic disorder
* Major gastrointestinal surgeries
* Patent ductus arteriosus (PDA) ligation surgery
* Outborn deliveries greater than 7 days old

Min Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Post menstrual Age (PMA) once full oral feeds are achieved as documented by not requiring gavage tube feeds for at least 24 hours | 2 months after enrollment
  Measured in the electronic medical record

SECONDARY OUTCOMES:
PMA at hospital discharge | up to 6 months after admission
PMA at completion of first oral feed | 1 month after enrollment.
length of hospitalization | up to 6 months after admission
number of gastrostomy tube | up to 6 months after admission
oxygen at discharge | up to 6 months after admission
safety outcomes during the feed as measured by the number of desaturations | 2 months after enrollment
safety outcomes during the feed as measured by the number of apnea episodes | 2 months after enrollment
safety outcomes during the feed as measured by the number of bradycardia episodes | 2 months after enrollment
safety outcomes as measured by the increase in fraction of inspired oxygen (FiO2) during and after feed | 2 months after enrollment
safety outcomes as measured by the increase in flow after feed | 2 months after enrollment
safety outcomes as measured by the number of choking episodes | 2 months after enrollment
safety outcomes as measured by the number of episodes of aspiration pneumonia | 2 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Ashley N Morin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No